CLINICAL TRIAL: NCT06503744
Title: Transthoracic Versus Transbronchial Ablation for Peripheral Lung Cancer Staging IA: a Prospective, Randomized Controlled Trial
Brief Title: Transthoracic vs Transbronchial Ablation for Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHCHE202301
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer Stage IA
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transthoracic ablation (Active Comparator): Transthoracic ablation
  Interventions: Procedure: ablation
- Transbronchial ablation (Experimental): Transbronchial ablation
  Interventions: Procedure: ablation

INTERVENTIONS:
Procedure: ablation — ablation

SUMMARY:
The aim of this study is to investigate the efficacy and safety of transthoracic versus transbronchial ablation in the treatment of early stage peripheral lung cancer.

DETAILED DESCRIPTION:
Ablation therapy has been widely used in the treatment of lung cancer and traditionally performed by CT-guided transthoracic puncture. In recent years, with the development of navigational bronchoscopy, exploratory studies on transbronchial ablation for peripheral lung cancer have demonstrated its efficacy and safety, but there is a lack of prospective randomized controlled trials to verify its near-term efficacy and safety, as well as its long-term efficacy. This study was designed as a prospective randomised controlled trial with 110 patients expected to participate in the study, randomized in a 1:1 ratio to CT-guided ablation and bronchoscopy-guided ablation treatment groups. The primary study endpoint is the rate of complete ablation at 6 months post-procedure. Secondary study endpoints were success rate of technique implementation, complete ablation rate at 12 months post-procedure, local control rate at 1, 2 and 3 years post-procedure, progression-free survival, overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years.
2. Primary peripheral lung cancer diagnosed by pathology and pre-procedure staging examination suggesting clinical stage T1N0M0, stage IA (including postoperative new and multiple primary).
3. The proposed ablation lesion was evaluated for feasibility of CT and bronchoscopy-guided ablation treatment.
4. Consent to initial ablation therapy is given after assessment of unsuitability for surgery or refusal of surgery and signed informed consent form.

Exclusion Criteria:

1. Patients with platelets <50×109/L, severe bleeding tendency and coagulation dysfunction that cannot be corrected in the short term.
2. Patients with severe pulmonary fibrosis and pulmonary arterial hypertension.
3. Infectious and radioactive inflammation around the lesion, skin infection at the puncture site that is not well controlled, systemic infection, high fever >38.5°C.
4. Patients with severe hepatic, renal, cardiac, pulmonary and cerebral insufficiency, severe anaemia, dehydration and serious disorders of nutritional metabolism that cannot be corrected or improved in the short term.
5. Those with poorly controlled malignant pleural effusions.
6. Anticoagulation therapy and/or anti-platelet drugs (except dabigatran, rivaroxaban and other new oral anticoagulants) have not been discontinued more than 5~7d before ablation.
7. Eastern Cooperative Oncology Group (ECOG) score >2.
8. Combination of other tumours with extensive metastases and an expected survival of <6 months.
9. Patients with episodic psychosis.
10. Patients with implanted electronic devices (e.g. pacemakers or defibrillators).
11. Pregnant women, or patients with a pregnancy planned during the study period.
12. Have participated or are participating in other clinical studies within the last 30 days.
13. Any other condition that the investigator considers inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate at 6 months post-procedure | Up to 6 months
  This refers to the number of lesions completely ablated 6 months after ablative treatment as a proportion of the total number of ablative treated lesions.

SECONDARY OUTCOMES:
Success rate of technique implementation | Immediate postoperative
  Defined as the number of lesions reached by the ablation needle and successfully treated by ablation as a proportion of the total number of lesions to be ablated, as assessed by imaging immediately after ablation.
Complete ablation rate at 12 months post-procedure | Up to 12 months
  This refers to the number of lesions completely ablated 12 months after ablative treatment as a proportion of the total number of ablative treated lesions.
Local control rate at 1, 2 and 3 years post-procedure | Up to 36 months
  This refers to the number of completely ablated and incompletely ablated lesions at 1, 2 and 3 years after ablative treatment as a proportion of the total number of ablative treated lesions.
Progression-free survival | Up to 36 months
  Refers to the duration between the subject's study procedure and the first occurrence of disease progression or death from any cause, recorded through follow-up for up to 3 years.
Overall survival | Up to 36 months
  Refers to the duration between the subject's study procedure and the subject's death, recorded through follow-up for up to 3 years.
Safety | Up to 6 months
  Assessment of the incidence of device or procedure-related adverse events that occurred during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, PhD, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China